CLINICAL TRIAL: NCT02632292
Title: EverolimuS-ElUtinG BioresorbAble VasculaR Scaffolds vErsus EVerolimus-Eluting Stents in Patients With Diabetes Mellitus
Acronym: SUGAR-EVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Luebeck (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); Kerckhoff Klinik (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Holger Thiele, Principal Investigator, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-260
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absorb GT1 (Experimental): Bioresorbable everolimus-eluting scaffolds
  Interventions: Device: Absorb GT1
- Promus (Active Comparator): Everolimus-eluting stents
  Interventions: Device: Promus

INTERVENTIONS:
Device: Absorb GT1 — Bioresorbable vascular scaffold
  Arms: Absorb GT1
Device: Promus — Everolimus-eluting stent
  Arms: Promus

SUMMARY:
Prospective, randomized, controlled, multicenter, open-label study to compare everolimus-eluting bioresorbable vascular scaffolds to everolimus-eluting stents in patients with diabetes mellitus.

ELIGIBILITY:
Clinical inclusion criteria:

* Age ≥18 years
* DM type I or II based on the definitions of the American Diabetes Association
* Angiographically proven CAD
* Angina pectoris, equivalent symptoms, and/or positive stress test, and/or instantaneous flow reserve ≤0.86, and/or fractional flow reserve ≤0.80
* Negative pregnancy test in women with childbearing potential

Angiographic inclusion criteria:

* De-novo lesion in at least one native coronary artery
* Luminal diameter reduction 50-99% assessed by visual estimation
* Target reference vessel diameter 2.5 - 4.0 mm

Clinical exclusion criteria:

* Limited long-term prognosis with a life-expectancy <12 months
* Contraindications to antiplatelet therapy
* Known allergy against cobalt chrome, everolimus, or polylactic acid

Angiographic exclusion criteria:

* Target lesion located in the left main trunk
* Severe calcification of the target lesion as determined by angiography
* In-stent restenosis
* Bifurcation lesion with planned two-stent strategy
* Chronic total occlusion
* Indication for CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss | Angiography 8-10 months after the index procedure

SECONDARY OUTCOMES:
Device success | Baseline angiography
  Attainment of <30% final residual stenosis following the index procedure.
Procedure success | Baseline angiography
  Device success and no periprocedural complications.
Vasomotion | Angiography 8-10 months after the index procedure
  Change in minimal lumen diameter before and after nitrate administration assessed by angiography at 8-10 months.
In-segment late lumen loss | Angiography 8-10 months after the index procedure
  Difference between the immediate post-procedure in-stent minimal lumen diameter and the in-stent minimal lumen diameter assessed by angiography at 8-10 months inside the stent or within 5 mm proximal or distal to the stent.
Binary restenosis | Angiography 8-10 months after the index procedure
  In-stent or in-segment restenosis ≥50% assessed by angiography at 8-10 months.
Conformability | Angiography 8-10 months after the index procedure
  Change in curvature and angulation between preprocedure, postprocedure, and angiographic follow-up at 8-10 months.
Major adverse cardiac events | 12- and 24-months
  Composite of cardiac death, myocardial infarction, scaffold/stent thrombosis, and target vessel revascularization
Cardiac death | 12- and 24-months
Myocardial infarction | 12- and 24-months
Scaffold/stent thrombosis | 12- and 24-months
Target vessel revascularization | 12- and 24-months
Target lesion failure | 12- and 24-months
  Composite of cardiac death, target vessel myocardial infarction and clinically driven target lesion revascularization
Target vessel failure | 12- and 24-months
  Composite of cardiac death, target vessel related myocardial infarction, clinically driven target vessel revascularization, and scaffold/stent thrombosis
Clinical success | 12- and 24-months
  Procedure success and no major adverse cardiac events at 12- and 24-month clinical follow-up
Anginal status assessed by the Seattle Angina Questionnaire | 12- and 24-months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Germany